CLINICAL TRIAL: NCT00710151
Title: Neurotoxicity in Primary Central Nervous System Lymphoma: An International, Collaborative, Observational Study of Cognition in Long-Term Survivors
Brief Title: Neurotoxicity in Primary Central Nervous System Lymphoma (PCNSL): An International Observational Study of Cognition in Long Term Survivors
Status: Terminated | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Other Study IDs: IRB00003805; R01NS033618 (NIH); OHSU-3805 (Other: OHSU IRB); NCT00706472 (obsolete NCT alias)
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL)
Keywords: neurotoxicity; cognition in survivors; diagnostic imaging
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Subjects with PCNSL who have survived disease-free for 2 years or more. Treatments will vary depending upon site of enrollment and will include chemotherapy, blood brain barrier disruption (BBBD) with chemotherapy, radiation, and stem cell transplantation.

SUMMARY:
This research is being done to investigate cognition in long term survivors of Primary Central Nervous System Lymphoma (PCNSL). Sometimes caregivers as well as patients who no longer have the disease report cognitive problems such as reduced memory or attentional dysfunction and decreased quality of life. Unfortunately, little is known about what may contribute to this cognitive dysfunction in part because PCNSL is a rare disease and sensitive tests have not often been used in the research studies. This project is being conducted to help understand what factors, such as radiation, may contribute to cognitive dysfunction and better define the relationship between brain structure and thinking in people who have had PCNSL.

DETAILED DESCRIPTION:
This is an international, multi-center project that will enroll as many as 118 subjects of which approximately 35 will be enrolled at Oregon Health & Science University (OHSU). Neuropsychological testing will consist of a battery of paper and pencil tests that examine abilities such as memory, motor skills, attention and speed of information processing. Questionnaires that assess quality of life will also be administered. These noninvasive tests are administered by a trained examiner or neuropsychologist and last about 30 minutes. Subjects will also undergo an MRI of the head which provides a picture of the brain's structure by placing an individual inside a powerful magnet. Statistical analyses will examine the relationship between the neuropsychological test scores and magnetic resonance (MR) images as well as examine the contribution of factors such as radiation, age, surgery, chemotherapy etc. to cognition.

ELIGIBILITY:
Inclusion Criteria:

* Radiological and histological diagnosis of PCNSL
* Age 18 years or older
* Survived 2 years or more following treatment
* Able to complete neuropsychological and neuroimaging parts of the study
* Signed a written informed consent in accordance with institutional guidelines

Exclusion Criteria:

* Subject has experienced recurrent disease
* Subject has a contraindication for MRI
* Subject has a contraindication for neuropsychological testing
* Subject has stage IV or V renal insufficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have had PCNSL and have survived disease-free for 2 years or more.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Neuropsychological Functioning | More than 2 years after treatment

SECONDARY OUTCOMES:
MRI | More than 2 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Neuwelt, MD, Principal Investigator — Oregon Health and Science University
Locations (4):
- Oregon Health & Science University, Portland, Oregon, United States
- Germany (3):
  - Charite University Medicine, Berlin
  - University of Bochum, Bochum
  - University Medical Center, Freiburg im Breisgau